CLINICAL TRIAL: NCT05746897
Title: A Phase 1 Study to Investigate the Safety, Tolerability, Pharmacokinetics/Pharmacodynamics, and Antitumor Activity of NM1F as Monotherapy and in Combination With Pembrolizumab in Subjects With Locally Advanced/Metastatic Solid Tumors
Brief Title: A First-in-human, Phase I, Open-label, Multicenter Study of NM1F(Anti-PVRIG) in Patients With Advanced Solid Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Hefei TG ImmunoPharma Co., Ltd. (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NM1F-T1-01
Record Dates: First submitted 2023-02-03; First posted 2023-02-28 (Actual); Last update posted 2024-01-26 (Actual); Status verified 2024-01

CONDITIONS: Ovarian Cancer; Melanoma; Triple Negative Breast Cancer; Colorectal Cancer
Keywords: solid tumors，NM1F，Pembrolizumab
MeSH Terms: conditions — Ovarian Neoplasms; Melanoma; Triple Negative Breast Neoplasms; Colorectal Neoplasms | interventions — pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- NM1F Injection/pembrolizumab Injection (Experimental): NM1F monotherapy dose escalation(Phase 1a) NM1F dose escalation in combination with a fixed dose of pembrolizumab(Phase 1b)
  Interventions: Drug: NM1F Injection; Drug: Pembrolizumab injection

INTERVENTIONS:
Drug: NM1F Injection — This is a Phase 1, multicenter, open-label, two-parts, FIH study to evaluate the tolerability, safety, PK/PD, and preliminary anti-tumor activity of NM1F as monotherapy and in combination with pembrolizumab (Keytruda®) in subjects with unresectable locally advanced, or metastatic solid tumors.
  The study consists of two parts: NM1F monotherapy dose escalation (Phase 1a), NM1F dose escalation in combination with a fixed dose of pembrolizumab (Phase 1b). For each subject in the two parts, the study will include a screening period (up to 28 days), a treatment period (until treatment discontinuation), and a follow-up period.
Drug: Pembrolizumab injection — This is a Phase 1, multicenter, open-label, two-parts, FIH study to evaluate the tolerability, safety, PK/PD, and preliminary anti-tumor activity of NM1F as monotherapy and in combination with pembrolizumab (Keytruda®) in subjects with unresectable locally advanced, or metastatic solid tumors.
  The study consists of two parts: NM1F monotherapy dose escalation (Phase 1a), NM1F dose escalation in combination with a fixed dose of pembrolizumab (Phase 1b). For each subject in the two parts, the study will include a screening period (up to 28 days), a treatment period (until treatment discontinuation), and a follow-up period.

SUMMARY:
A Phase 1 Study to Investigate the Safety, Tolerability, Pharmacokinetics/Pharmacodynamics, and Antitumor Activity of NM1F as Monotherapy and in Combination with Pembrolizumab in Subjects with Locally Advanced/Metastatic Solid Tumors

DETAILED DESCRIPTION:
This is a Phase 1, multicenter, open-label, two-parts, FIH study to evaluate the tolerability, safety, PK/PD, and preliminary anti-tumor activity of NM1F as monotherapy and in combination with pembrolizumab (Keytruda®) in subjects with unresectable locally advanced, or metastatic solid tumors.

The study consists of two parts : NM1F monotherapy dose escalation (Phase 1a), NM1F dose escalation in combination with a fixed dose of pembrolizumab (Phase 1b). For each subject in the two parts, the study will include a screening period (up to 28 days), a treatment period (1 year and 2 years for Phase 1a and 1b, respectively, or until treatment discontinuation), and a follow-up period .

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects age ≥ 18 years at the time of informed consent.
2. Subjects with histologically or cytologically diagnosed unresectable locally advanced, or metastatic solid tumors, mainly but not limited to CRC, TNBC, melanoma, OC, and who have progressed despite all standard therapy or are intolerant of all standard therapy, or for whom no effective standard therapy exists
3. Subjects must have at least 1 evaluable lesion as defined by response evaluation criteria in solid tumors (RECIST) v1.1.
4. ECOG PS of 0~2.
5. Life expectancy ≥ 3 months.
6. Subjects have sufficient baseline organ function and laboratory data.
7. Woman of childbearing potential must have a negative serum pregnancy test within 7 days prior to treatment.
8. Female subjects of childbearing potential or male subjects with a partner of childbearing potential must agree to use effective contraception at the time of informed consent and continuing through the study until 6 months after the last dose of NM1F and / or pembrolizumab.

   -

Exclusion Criteria:

Cancer Related

1. Subject with known active central nervous system (CNS) primary tumor or metastases.
2. History of intercurrent severe chronic or active infections.
3. Has a history of active autoimmune diseases , or is receiving chronic systemic steroid therapy (in dosing exceeding 10 mg daily of prednisone equivalent) or any other form of immunosuppressive therapy within 14 days prior the first dose of study drug.
4. Has a history of symptomatic interstitial lung disease or inflammatory pneumonitis.
5. Has a history of impaired cardiac function or clinically significant cardiovascular diseases.
6. Prior allogenic or autologous bone marrow transplantation or other solid organ transplantation.
7. Has a known additional malignancy that is progressing or has required active treatment within the past 3 years (Note: Exceptions are subjects with basal cell carcinoma of the skin, squamous cell carcinoma of the skin, and localized prostate cancer who have undergone potentially curative therapy. These subjects are not excluded).
8. Evidence of clinically significant immunosuppression such as the following:

   1. Primary immunodeficiency state such as Severe Combined Immunodeficiency Disease (SCID)
   2. Concurrent opportunistic infection
9. Presence of uncontrolled pleural effusion, pericardial effusion or ascites requiring recurrent drainage procedures (monthly or more frequently).
10. Has received prior anticancer treatment with the following therapies (specified time periods are from last dose of prior treatment to first dose of NM1F):

    1. Any therapy directed against PVRIG (COM701 or other anti-PVRIG mAb) or other CD226 axis receptor (TIGIT or CD96) at any time.
    2. Chemotherapy, target therapy, immunotherapy, or other anticancer therapy within 28 days or 5 half-lives, whichever is shorter, prior to the first dose of study treatment.
    3. Prior radiotherapy ≤ 4 weeks prior to the first dose of study treatment, with the exception of a single fraction of radiotherapy for the purposes of palliation, which is permitted.
    4. Investigational therapy: if the subject has participated in a clinical study and has received an investigational product within 4 weeks prior to the first dose of study treatment.
11. Has received systematic immunomodulatory drugs within 14 days before the first dose of study drug, such as thymosin, IL-2, IFN.
12. Has received a live vaccine within 4 weeks prior to the first dose of study drug.
13. Has a recent major surgery within 4 weeks prior to the first dose of study drug or is expected to undergo major surgery during the study.
14. Toxicities of prior therapies have not been resolved to ≤ Grade 1 or baseline as per NCI-CTCAE v5.0, except for alopecia, skin hyperpigmentation.
15. Subjects who have experienced Grade ≥ 3 irAEs from prior immunotherapies or who discontinue immunotherapy due to immune-related toxicities.
16. Has a known psychiatric or substance abuse disorder that would interfere with the subject's ability to cooperate with the requirements of the study.
17. Pregnancy or lactation. Women who are willing to discontinue breastfeeding prior to administration of study drug and do not intend to resume breastfeeding may be enrolled.
18. Has known hypersensitivity to either the drug substances or inactive ingredients in the drug product.
19. Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the study, interfere with the subject's participation for the full duration of the study, or is not in the best interest of the subject to participate, in the opinion of the investigator.
20. Subjects who are unwilling or unable to comply with study procedures and study restrictions, or in the judgment of the investigator, would make the subject inappropriate for entry into this study.
21. Subjects who have contraindication for use of PD-1/PD-L1 antibody (only for Phase 1b).

    -

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Estimated)
Dates: Start 2023-04-13 (Actual); Primary Completion 2027-09-30 (Estimated); Study Completion 2027-09-30 (Estimated)

PRIMARY OUTCOMES:
Dose-limiting Toxicity (DLT) | First 21 days of treatment.
  The incidence of DLTs during the DLT assessment period.
Dose-Finding | Approximately 3 years.
  Determination of the MTD or maximum tested dose, and the RP2D.
Frequency and Severity of Adverse Events (AE) | Screening to 30 days from last dose
  The incidences and percentages of patients experiencing AEs summarized by NCI CTCAE version 5.0 grade and by causality.

SECONDARY OUTCOMES:
Pharmacokinetics of NM1F | Day 1 of dosing through 30 days post last dose
  Maximum Plasma Concentration (Cmax)
Pharmacokinetics of NM1F | Day 1 of dosing through 30 days post last dose
  Area Under the Curve (AUC)
Number of subjects with Anti-NM1F antibody positive . | Day 1 of dosing through 30 days post last dose
  Immunogenicity of NM1F monotherapy and in combination with pembrolizumab
Objective Response Rate (ORR) | Approximately 3 years.
  ORR according to RECIST v1.1.
Duration of Response (DoR) | Approximately 3 years.
  Time from the date measurement criteria are first met for PR or CR to the date measurement criteria are first met for progressive disease.
Disease Control Rate (DCR) | Approximately 3 years.
  The proportion of subjects who have best overall response of CR or PR, or stable disease (SD).
Progression Free Survival (PFS) | Approximately 3 years.
  Time from the date of initiation of study therapy to the date measurement criteria are first met for progressive disease or death from any cause, whichever occurs first.
Overall Survival (OS) | Approximately 3 years.
  Time from the date of initiation of study therapy to the date of death from any cause.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - NEXT Oncology, Dallas, Dallas, Texas
  - Next Oncology, Virginia Cancer Specialists, Fairfax, Virginia

IPD SHARING:
Plan to Share IPD: No